CLINICAL TRIAL: NCT02639169
Title: The Impact of Music Therapy on Mood Control in Hospitalized Patients for Transplantation of Hematopoietic Stem Cells
Brief Title: Music Therapy Improves the Mood of Patients Undergoing Hematopoietic Stem Cells Transplantation
Acronym: MTHSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Carlos Antonio Dóro, Principal Investigator, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 26404414.9.0000.0096
Record Dates: First submitted 2015-12-10; First posted 2015-12-24 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Mood
Keywords: music therapy; Distress; Mood; HSCT
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- music (Experimental): Apply live music through techniques music therapy in group experimental and evaluation through the visual analog scale (VAS) and numeric.
  Interventions: Other: Music Therapy
- Comparative (No Intervention): Apply the visual analog scale (VAS) and numeric.

INTERVENTIONS:
Other: Music Therapy — apply live music through the techniques of music therapy
  Arms: music

SUMMARY:
ABSTRACT The transplant allogeneic hematopoietic stem cell transplantation (HSCT Alo) is a therapeutic medical treatment carried out in combat various neoplastic hematologic disorders, congenital, genetic or acquired. In this procedure, which combines high-dose chemotherapy and or radiation and has a degree of high cytotoxicity, the patient goes for a social solitary confinement, which causes psychological distress, pain, anxiety, mood disorders and can lead to depression. The music therapy was applied and the purpose of decreasing the insulation. This is a randomized controlled study.

Method: Apply the intervention of live music sessions through the techniques of music therapy; assess and quantify through the visual analog scale (VAS) and numeric. The dependent variables, pain, anxiety and mood of the participants selected randomly for the experimental group music therapy (EGM) n=50, and compare with the control group (CG) n=50, which received only the standard treatment.

DETAILED DESCRIPTION:
METHODOLOGY Study Design. It is a randomized controlled experimental study Place: Clinical Hospital Complex of the Federal University of Parana, Bone Marrow Transplant Service. The research was developed in the period Jan/2014 to November/2015.

Population: Adult patients undergoing hematopoietic stem cell transplantation (HSCT) Allogeneic. Approved by the Ethics Committee in Research of the University Federal of Paraná Clinical Hospital Complex, Presentation certificate for consideration Ethics: 26404414.9.0000.0096 Sample Calculation: The calculation of sample size was based on a previous pilot study for which was identified an average of 5.4 for the score of humor with standard deviation of 1.9. It was felt that this group corresponds to the control group of the new study and a minimal difference in the score of humor 1 point higher in the experimental group would be clinically relevant. For a significance level of 5% and a 80% test power, would take at least 45 cases in each group (Control and Experimental). Depending on the evaluation of mood score is given by an ordinal scale, it is suggested a 10% increase in the sample size in each group. Thus, 50 patients were needed in each group. the calculation of the sample was done by statistical.

Randomization: It was made random and concealed allocation of participants in the groups as follows: A Contributor not involved with the research played a given and communicated the number randomly selected to the researcher, the number was pair, and would compose the experimental group of music therapy. If it was odd participant would make up the control group. The evaluation was done by an external student of psychology. For musical intervention was not possible to apply the principle of double blind but, the evaluator did not know what kind of intervention was applied. The interventions were applied twice a week on Tuesdays and Thursdays from 9:00 am to 12:00 pm. in the morning and the assessment on the same day but the afternoon.

METHOD Apply live music through the music therapy techniques such as re-creation, improvisation and rhythmic production, the experimental group of music therapy (EGM).

Implement and measure through the visual analog scale (VAS) and numeric the level of mood, anxiety and pain in the experimental group music therapy (EGM).

Apply the visual analog scale (VAS) and numeric to measure the levels of Mood, Anxiety and Pain Control Group (GC) that received only the standard treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* The invitation was made to each patient submitted to (HSCT Alo) with aged between 18 and 65 years.
* If the patient accepted to participate in the research should sign a free and informed consent form (ICF)

EXCLUSION CRITERIA:

* All patients who did not undergoing allogeneic transplantation were excluded also in case of opting out of the search
* All minors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mood | "1 year"
  The Mann Whitney test Showed statistical of significance p <0.05

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Doro, Student, Principal Investigator — Universidade Federal do Parana

IPD SHARING:
Plan to Share IPD: Yes
Result of data collected during the research in tables calculated by a statistical

REFERENCES:
- [Background] BRUSCIA K. E. Definindo a Musicoterapia. Rio de Janeiro, Ed. Enelivros - 2000.
- [Background] Jacobsen PB, Donovan KA, Trask PC, Fleishman SB, Zabora J, Baker F, Holland JC. Screening for psychologic distress in ambulatory cancer patients. Cancer. 2005 Apr 1;103(7):1494-502. doi: 10.1002/cncr.20940. PMID 15726544
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] MACHADO, L.N; CAMANDONI, V.O; HARO LEAL K.P; MOSCATELLO, E.L.M. Transplante de Medula Óssea Abordagem Multidisciplinar São Paulo Lemar 2009
- [Background] ORTEGA, E.T.T; KOJO, T.K; DE LIMA, D.H; VERAN, M.P; NEVES, M. I. Compêndio de Enfermagem em Transplante de Células-Tronco Hematopoéticas Editora Maio Curitiba 2004
- [Background] PETERSEN, E.M; Revista do Hospital Universitario Pedro Ernesto UERJ - 2012
- [Result] Bradt J, Dileo C, Grocke D, Magill L. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD006911. doi: 10.1002/14651858.CD006911.pub2. PMID 21833957
- [Result] Ratcliff CG, Prinsloo S, Richardson M, Baynham-Fletcher L, Lee R, Chaoul A, Cohen MZ, de Lima M, Cohen L. Music therapy for patients who have undergone hematopoietic stem cell transplant. Evid Based Complement Alternat Med. 2014;2014:742941. doi: 10.1155/2014/742941. Epub 2014 Jan 9. PMID 24527052
- [Result] Raglio A, Attardo L, Gontero G, Rollino S, Groppo E, Granieri E. Effects of music and music therapy on mood in neurological patients. World J Psychiatry. 2015 Mar 22;5(1):68-78. doi: 10.5498/wjp.v5.i1.68. PMID 25815256